CLINICAL TRIAL: NCT07114861
Title: An Open-label, Dose-finding and Dose-expansion, Phase I/IIa Clinical Trial to Evaluate the Safety and Efficacy of KN510713 in Combination With mFOLFIRINOX in Patients With Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: The KN510713 Study in Combination With mFOLFIRINOX
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New Cancer Cure-Bio Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCCKN-101-P2a
Record Dates: First submitted 2025-07-23; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced or Metastatic Pancreatic Ductal Adenocarcinoma (PDAC)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KN510 120mg + KN713 90mg (Experimental)
  Interventions: Drug: Study drug: KN510 120mg/day + KN713 90mg/day, Combination Chemotherapy: mFOLFIRINOX
- KN510 120mg + KN713 120mg (Experimental)
  Interventions: Drug: Study drug: KN510 120mg/day + KN713 120mg/day, Combination Chemotherapy: mFOLFIRINOX

INTERVENTIONS:
Drug: Study drug: KN510 120mg/day + KN713 90mg/day, Combination Chemotherapy: mFOLFIRINOX — KN510 120mg/day + KN713 90mg/day: once daily in 14-day (2-week) cycles. mFOLFIRINOX: Treatment is repeated every 2 weeks
  Arms: KN510 120mg + KN713 90mg
Drug: Study drug: KN510 120mg/day + KN713 120mg/day, Combination Chemotherapy: mFOLFIRINOX — KN510 120mg/day + KN713 120mg/day: once daily in 14-day (2-week) cycles. mFOLFIRINOX: Treatment is repeated every 2 weeks
  Arms: KN510 120mg + KN713 120mg

SUMMARY:
This study is designed to evaluate the safety and efficacy of KN510713 in combination with mFOLFIRINOX in patients with locally advanced or metastatic pancreatic cancer. The study will be conducted in two parts: Part 1 (Dose-finding) and Part 2 (Dose expansion).

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female subjects aged 19 to 75 years at the time of providing written informed consent
2. Subjects with histologically or cytologically confirmed unresectable, locally advanced or metastatic PDAC who are scheduled to receive treatement with mFOLFIRINOX
3. Subjects who have not received prior systemic chemotherapy for locally advanced or metastatic pancreatic cancer (Note: Prior neo-adjuvant or adjuvant systemic chemotherapy is allowed if there was no disease progression within 6 months after the last dose of chemotherapy)
4. Subjects with at least one measurable lesion according to RECIST ver1.1
5. Subjects with an ECOG performance status of 0 or 1
6. Subjects with an expected survival of at least 12 weeks
7. Subjects with adequate hematologic function, renal and hepatic function, and coagulation function based on the following laboratory criteria (only one repeat of laboratory tests is permitted during the screening period)
8. Subjects who have been informed about the clinical study and voluntarily signed the written informed consent form

Exclusion Criteria:

1) Known hypersensitivity to the IP, combination anticancer agents, their components, or drugs of a similar class 2) Subjects with any of the following medical history, or surgical/procedural history identified:

1. History of any malignancy other than pancreatic cancer within 5 years prior to screening (Subjects with a history of basal cell carcinoma, squamous cell carcinoma of the skin, thyroid cancer, or carcinoma in situ at other sites may be eligible if the cancer was successfully treated and there has been no recurrence for more than 3 years, as determined by the investigator).
2. Major surgery requiring general anesthesia or ventilatory support within 4 weeks prior to baseline (Video-assisted thoracoscopic surgery (VATS) or ONC surgery is limited to 2 weeks).
3. Clinically significant arrhythmia, acute myocardial infarction, unstable angina, or NYHA class III or IV heart failure within 24 weeks prior to baseline.
4. Pulmonary thrombosis, deep vein thrombosis, or other serious, life-threatening pulmonary diseases (e.g., acute respiratory distress syndrome, lung failure), or conditions such as asthma or COPD considered inappropriate for study participation, occurring within 24 weeks prior to baseline.
5. Known DPD deficiency
6. Subjects known to carry the genetic polymorphism of UGT1A1*6 or UGT1A1*28 as homozygotes (UGT1A1*6/*6 or UGT1A1*28/*28) or as compound heterozygotes (UGT1A1*6/*28)
7. Known fructose intolerance 3) Comorbidities or conditions as follows:

(1) Peripheral neuropathy of moderate (Grade 2) or higher (2) Chronic diarrhea or inflammatory bowel disease (Crohn's disease, ulcerative colitis) (3) Ileus or Intestinal obstruction (4) Clinically significant symptoms of ILD or pulmonary fibrosis requiring steroid therapy (5) Chronic kidney disease requiring dialysis (6) Clinically significant symptomatic or uncontrolled central nervous system or brain metastases (permitted if systemic corticosteroids were discontinued ≥4 weeks prior to baseline and the metastases have remained stable for ≥4 weeks) (7) Uncontrolled hypertension (SBP/DBP ≥160/100 mmHg) (8) QTc >450 ms on ECG (9) Active hepatitis B or hepatitis C (10) Known HIV infection (11) Conditions interfering with oral intake (e.g., dysphagia) or absorption (e.g., celiac disease, Crohn's disease, or a clinically significant bowel resection that may affect drug absorption) (12) Subjects with a history or suspected symptoms of gastro-esophageal reflux disease (GERD), including gastric ulcer, duodenal ulcer, or reflux esophagitis (13) Parkinson's disease, parkinsonism, tremor, restless leg syndrome, or other related movement disorders (14) Clinically significant symptomatic or uncontrolled ascites or pleural effusion (15) Subjects who, in the investigator's judgment, have a disease or condition sufficiently serious to influence the study results, or for whom the concomitant anticancer agents are contraindicated 4) Prior medications or treatments as follows:

1. Radiotherapy within 2 weeks prior to screening (radiotherapy for symptom relief or bone lesions at high risk of pathological fracture is allowed if completed ≥1 week before the planned enrollment, provided that the treated lesions is not selected as target lesions for RECIST evaluation)
2. Use of PPIs other than the IP within 2 weeks prior to screening
3. Administration of any antithrombotic agents, including antiplatelet or anticoagulant drugs, within 2 weeks prior to screening, or an anticipated need for such medication during the study period (the use of low-molecular-weight heparin [LMWH] for prophylaxis or management of venous thrombosis is permitted during the study)
4. Use of rilpivirine-containing products within 2 weeks prior to screening
5. Use of atazanavir-containing products within 2 weeks prior to screening
6. Current administration of, or anticipated need for strong CYP3A4 inhibitors or inducers
7. Current administration of, or anticipated need for CYP2C19 substrates, strong inhibitors, or inducers
8. High dose methotrexate (≥1000 mg/m2)
9. St. John's wort
10. Requirement for continuous use (≥4 weeks) of systemic corticosteroids equivalent to >10 mg/day prednisone (local administration such as intra-articular, intranasal, ophthalmic, or inhaled corticosteroids, and short-term use for the treatment or prophylaxis of contrast-media allergy or AEs [e.g., vomiting] are permitted)
11. Current administration of, or anticipated need for sorivudine 5) Pregnant or breastfeeding women, or women of childbearing potential and men who are unwilling to remain abstinent or use appropriate contraception until 12 months (for men) or 15 months (for women) after the last administration of IP/concomitant medication following study enrollment 6) Participation in another clinical trial and administration or application of an investigational drug or device within 4 weeks prior to screening 7) Any other subject who, in the investigator's judgment, is unsuitable for participation in this study

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-22 (Estimated); Primary Completion 2028-09-22 (Estimated); Study Completion 2028-10-22 (Estimated)

PRIMARY OUTCOMES:
Number of occurrences, affected subjects with adverse events. | Through study completion, an average of 12 months
  Safety Evaluation(Adverse Event, Laboratory Test, Vital Signs, Electrocardiogram)
The frequency and percentage of Dose-Limiting Toxicitys | 4 weeks
  Safety/Tolerability Evaluation(Dose-Limiting Toxicity, Part 1 Subjects only)

SECONDARY OUTCOMES:
Objective Response Rate | Through study completion, an average of 12 months
  The proportion of subjects whose best overall response (BOR) is assessed as complete response (CR) or partial response (PR). ORR = CR + PR
Disease Control Rate | Through study completion, an average of 12 months
  The proportion of subjects whose BOR is assessed as CR, PR, or stable disease (SD). DCR = CR + PR + SD
Duration of Response | Through study completion, an average of 12 months
  The duration from the date of the first assessment of CR or PR to the date of the first assessment disease progression (PD)
Progression-Free Survival | Through study completion, an average of 12 months
  The time from the start date of IP administration to the earlier of either PD based on RECIST ver1.1 or death from any cause
Overall Survival | Through study completion, an average of 12 months
  The time from the start date of IP administration to the date of death from any cause

OTHER OUTCOMES:
Changes in Phospholipids | Screening, 8 weeks
  The number of subjects, mean, standard deviation, median, minimum, and maximum will be presented for changes at each time point.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang-si, South Korea